CLINICAL TRIAL: NCT00603668
Title: A Phase I/II Study of Immunotherapy With Milatuzumab (hLL1) in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Phase I/II Study of Different Doses and Dose Schedules of Milatuzumab (hLL1) in CLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hLL1-02
Record Dates: First submitted 2008-01-08; First posted 2008-01-29 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2013-03

CONDITIONS: Chronic Lymphocytic Lymphoma
Keywords: CLL
MeSH Terms: interventions — milatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- milatuzumab (Experimental): different doses of hLL1
  Interventions: Biological: milatuzumab

INTERVENTIONS:
Biological: milatuzumab — two or three times a week dosing of hLL1 for a total of 4 weeks
  Other Names: IMMU-115; hLL1

SUMMARY:
This study will test different doses of anti-CD74 antibody in patients with NHL and/or CLL.

DETAILED DESCRIPTION:
Milatuzumab (hLL1, IMMU-115), a humanized anti-CD74 monoclonal antibody. Dose escalation will utilize 4 planned dose regimens with 4.0 or 8.0 mg/kg doses administered intravenously either twice weekly (days 1 and 4) or thrice weekly (days 1, 3 and 5) for 4 consecutive weeks. The four planned dose regimens will be labeled as dose level 1 to 4 corresponding to increasing levels of the total dose of milatuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of recurrent chronic lymphocytic leukemia (by NCI criteria)
* Received at least one prior treatment with standard therapy (previous antibody therapy is acceptable)
* Measurable disease (WBC > 5,000 for CLL)
* See protocol for full list

Exclusion Criteria:

* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control while enrolled in the study until at least 12 weeks after the last milatuzumab infusion
* Prior therapy with other human or humanized monoclonal antibodies, unless HAHA tested and negative;
* Bulky disease by CT, defined as any single mass >10 cm in its greatest diameter
* Known HIV positive or active hepatitis B or C, or presence of hepatitis B surface antigens or presence of hepatitis C antibody
* Known autoimmune disease or presence of autoimmune phenomena
* At least 7 days beyond any infection requiring antibiotic use.
* Systemic corticosteroids within 2 weeks, except low dose regimens (prednisone, <20 mg/day, or equivalent) which may continue if unchanged.
* Substance abuse or other concurrent medical or psychiatric conditions that, in the Investigator's opinion, could confound study interpretation or affect the patient's ability to tolerate or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety of the anti-CD74 antibody will be evaluated based upon physical examinations, hematology and chemistry laboratory evaluations and toxicity events | over first 12 weeks

SECONDARY OUTCOMES:
Efficacy (to see if the study drug works) in patients with NHL and CLL | over the first 12 weeks, then over up to 2 years
Pharmacokinetics (how the drug is processed by the body) | over the first 12 weeks
Pharmacodynamics (how the study drug is absorbed by the body)' | over the first 12 weeks, then over 2 years
Immunogenicity | over at least first 12 weeks
optimal dose | first 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (5):
- United States (5):
  - Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Georgetown University Hospital Lombardi Cancer Center, Washington D.C., District of Columbia
  - M. D. Anderson Cancer Center, Orlando, Florida
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Stein R, Mattes MJ, Cardillo TM, Hansen HJ, Chang CH, Burton J, Govindan S, Goldenberg DM. CD74: a new candidate target for the immunotherapy of B-cell neoplasms. Clin Cancer Res. 2007 Sep 15;13(18 Pt 2):5556s-5563s. doi: 10.1158/1078-0432.CCR-07-1167. PMID 17875789
- [Background] Stein R, Qu Z, Cardillo TM, Chen S, Rosario A, Horak ID, Hansen HJ, Goldenberg DM. Antiproliferative activity of a humanized anti-CD74 monoclonal antibody, hLL1, on B-cell malignancies. Blood. 2004 Dec 1;104(12):3705-11. doi: 10.1182/blood-2004-03-0890. Epub 2004 Aug 5. PMID 15297317